CLINICAL TRIAL: NCT01457586
Title: Observational Study of Hemoderivative Imputable Complications in Initial Uncomplicated Heart Surgery
Brief Title: Hemoderivative Imputable Complications in Initial Uncomplicated Heart Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Pitangueiras (Other)
Responsible Party: Principal Investigator, Roberto Rocha e Silva, MD PHD in Cardiac Surgery, Hospital Pitangueiras
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Heart surgery hemoderivatives
Record Dates: First submitted 2011-10-19; First posted 2011-10-24 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Heart Diseases
Keywords: Heart Surgery; Blood Transfusion; Postoperative Complications
MeSH Terms: conditions — Heart Diseases; Postoperative Complications | interventions — Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transfusion (Active Comparator): Patient who received blood transfusion in the perioperative period
  Interventions: Biological: Blood transfusion
- No Transfusion (No Intervention): Patients who did not receive blood transfusion in the perioperative period
  Interventions: Biological: No blood transfusion

INTERVENTIONS:
Biological: Blood transfusion — Blood transfusion in perioperative period.
  Arms: Transfusion
Biological: No blood transfusion — No transfusion in the perioperative period.
  Arms: No Transfusion

SUMMARY:
Observational Study of Hemoderivative Transfusion Imputable Complications in Initial Uncomplicated Heart Surgery. Inclusion criteria are patients who discontinued the mechanical ventilation up to 6 hours after exiting operation room and who discontinued vasoactive drugs up to the beginning of the second postoperative day.

Blood transfusion might be only a marker of the patient severity.

DETAILED DESCRIPTION:
Criteria for blood transfusion during extra corporeal circulation (if used) is volume expansion need leading to a predictable hematocrit lower than 25%.

Criteria for blood transfusion after extra corporeal circulation or in the postoperative period is a hematocrit below 30% with signs of low cardiac output due to hypovolemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acquired heart disease with indication for surgery and who discontinued the mechanical ventilation up to 6 hours after exiting operation room and who discontinued vasoactive drugs up to the beginning of the second postoperative day.

Exclusion Criteria:

* Patients who received blood transfusion previous to the heart surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Any postoperative complication | 1 month
  Postoperative complication up to 1 month. Comparison between patients who did or did not receive blood transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: ROBERTO R Silva, MD PHD, Principal Investigator — Hospital Pitangueiras
Locations (1):
- Hospital Pitangueiras, Jundiaí, São Paulo, Brazil

REFERENCES:
- [Background] Ranucci M, Pavesi M, Mazza E, Bertucci C, Frigiola A, Menicanti L, Ditta A, Boncilli A, Conti D. Risk factors for renal dysfunction after coronary surgery: the role of cardiopulmonary bypass technique. Perfusion. 1994;9(5):319-26. doi: 10.1177/026765919400900503. PMID 7833539
- [Background] Leal-Noval SR, Marquez-Vacaro JA, Garcia-Curiel A, Camacho-Larana P, Rincon-Ferrari MD, Ordonez-Fernandez A, Flores-Cordero JM, Loscertales-Abril J. Nosocomial pneumonia in patients undergoing heart surgery. Crit Care Med. 2000 Apr;28(4):935-40. doi: 10.1097/00003246-200004000-00004. PMID 10809262
- [Background] Zacharias A, Habib RH. Factors predisposing to median sternotomy complications. Deep vs superficial infection. Chest. 1996 Nov;110(5):1173-8. doi: 10.1378/chest.110.5.1173. PMID 8915216
- [Background] Michalopoulos A, Stavridis G, Geroulanos S. Severe sepsis in cardiac surgical patients. Eur J Surg. 1998 Mar;164(3):217-22. doi: 10.1080/110241598750004670. PMID 9562283
- [Background] Michalopoulos A, Tzelepis G, Dafni U, Geroulanos S. Determinants of hospital mortality after coronary artery bypass grafting. Chest. 1999 Jun;115(6):1598-603. doi: 10.1378/chest.115.6.1598. PMID 10378555
- [Background] Engoren MC, Habib RH, Zacharias A, Schwann TA, Riordan CJ, Durham SJ. Effect of blood transfusion on long-term survival after cardiac operation. Ann Thorac Surg. 2002 Oct;74(4):1180-6. doi: 10.1016/s0003-4975(02)03766-9. PMID 12400765
- [Background] Hung M, Besser M, Sharples LD, Nair SK, Klein AA. The prevalence and association with transfusion, intensive care unit stay and mortality of pre-operative anaemia in a cohort of cardiac surgery patients. Anaesthesia. 2011 Sep;66(9):812-8. doi: 10.1111/j.1365-2044.2011.06819.x. Epub 2011 Jul 25. PMID 21790520
- [Background] Dardashti A, Ederoth P, Algotsson L, Bronden B, Luhrs C, Bjursten H. Blood transfusion after cardiac surgery: is it the patient or the transfusion that carries the risk? Acta Anaesthesiol Scand. 2011 Sep;55(8):952-61. doi: 10.1111/j.1399-6576.2011.02445.x. Epub 2011 May 16. PMID 21574966